CLINICAL TRIAL: NCT02112227
Title: Patient-centered Care Transitions in Heart Failure: A Pragmatic Cluster
Brief Title: Patient-centered Care Transitions in Heart Failure: A Pragmatic Cluster Randomized Trial
Acronym: PACT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Harriette Van Spall, Assistant Professor of Medicine, Division of Cardiology, McMaster University, Population Health Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: PACT-HF
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Transitional Care; Knowledge Translation; Outcomes
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Discharge planning services (Active Comparator): Proven effective discharge-planning services will be grouped into 'patient-centered care transitions in heart failure' patients. This will be known as the PACT-HF model.
  Interventions: Other: PACT-HF Model
- Standard Care (No Intervention): Standard of care will be provided to HF patients at discharge.

INTERVENTIONS:
Other: PACT-HF Model — PACT-HF Model includes the following 1) comprehensive patient assessment 2) self-care education 3) patient-centered discharge summary 4) early follow up with FP 5) referral of high-risk patients to regional multidisciplinary HF clinic and to nurse-led home care
  Arms: Discharge planning services

SUMMARY:
Heart failure (HF) is the most common cause of hospitalization in older adults. The month after hospital discharge represents a vulnerable period, when patients are at increased risk of death and readmission to hospital. Research has shown that certain discharge-planning services can reduce death and readmissions, but these have not been widely implemented. In this study, we will group evidence-informed discharge-planning services into 'Patient-centered Care Transitions in HF' (PACT-HF), a model of care that will prepare patients for their transition from hospital to home. Through PACT-HF, patients will benefit from a comprehensive assessment of their health care needs, learn to recognize and manage symptoms of HF, and receive the information and follow-up care needed to optimize their health. We will introduce PACT-HF to 10 Ontario hospitals over a number of time periods using a stepped wedge cluster trial design. We will compare the outcomes (hierarchically ordered) of patients in hospitals with PACT-HF to those in hospitals without PACT-HF. We anticipate that patients hospitalized at the sites with PACT-HF will have fewer readmissions, emergency visits, and deaths after discharge; report a better quality of life; and feel more prepared for discharge. We also anticipate that overall, PACT-HF will reduce health system costs.

ELIGIBILITY:
Inclusion Criteria:

* In participating hospitals, all patients hospitalized with the most responsible diagnosis of Heart Failure

Exclusion Criteria:

* Patients who die during hospitalization or are transferred to another hospital

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Time to composite all-cause readmissions/emergency department (ED) visits/death at 3 months | Within 3 months of hospital discharge
Time to composite all-cause readmissions/emergency department (ED) visits/death at 30 days | Within 30 days of hospital discharge

SECONDARY OUTCOMES:
Preparedness for discharge | On admission, at 6 weeks and 6 months post discharge
  Patient-centered outcome, as measured by a validated survey instrument
Quality of life, as measured by the EQ5D5L scale | Administered on admission for HF and also 6 weeks and 6 months post discharge
  Health-related quality of life, as measured by the validated EQ5D5L scale. This will be administered on admission and within 6 weeks and 6 months of the patient's discharge.
Health Care Costs | 6 months post discharge
  Total health care system costs per patient, using the viewpoint of the Ministry of Health. This will be measured using administrative databases.

CONTACTS AND LOCATIONS:
Overall Officials: Harriette Van Spall, MD, Principal Investigator — McMaster University
Locations (1):
- Population Health Research Institute of McMaster University and Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Averbuch T, Lee SF, Zagorski B, Pandey A, Petrie MC, Biering-Sorensen T, Xie F, Van Spall HGC. Long-term clinical outcomes and healthcare resource utilization in male and female patients following hospitalization for heart failure. Eur J Heart Fail. 2025 Feb;27(2):377-387. doi: 10.1002/ejhf.3499. Epub 2024 Nov 5. PMID 39498574
- [Derived] Averbuch T, Lee SF, Zagorski B, Mebazaa A, Fonarow GC, Thabane L, Van Spall HGC. Effect of a transitional care model following hospitalization for heart failure: 3-year outcomes of the Patient-Centered Care Transitions in Heart Failure (PACT-HF) randomized controlled trial. Eur J Heart Fail. 2024 Mar;26(3):652-660. doi: 10.1002/ejhf.3134. Epub 2024 Feb 1. PMID 38303550
- [Derived] Van Spall HGC, DeFilippis EM, Lee SF, Oz UE, Perez R, Healey JS, Allen LA, Voors AA, Ko DT, Thabane L, Connolly SJ. Sex-Specific Clinical Outcomes of the PACT-HF Randomized Trial. Circ Heart Fail. 2021 Nov;14(11):e008548. doi: 10.1161/CIRCHEARTFAILURE.121.008548. Epub 2021 Oct 29. PMID 34711072
- [Derived] Blumer V, Gayowsky A, Xie F, Greene SJ, Graham MM, Ezekowitz JA, Perez R, Ko DT, Thabane L, Zannad F, Van Spall HGC. Effect of patient-centered transitional care services on patient-reported outcomes in heart failure: sex-specific analysis of the PACT-HF randomized controlled trial. Eur J Heart Fail. 2021 Sep;23(9):1488-1498. doi: 10.1002/ejhf.2312. Epub 2021 Aug 16. PMID 34302417
- [Derived] Gevaert AB, Tibebu S, Mamas MA, Ravindra NG, Lee SF, Ahmad T, Ko DT, Januzzi JL Jr, Van Spall HGC. Clinical phenogroups are more effective than left ventricular ejection fraction categories in stratifying heart failure outcomes. ESC Heart Fail. 2021 Aug;8(4):2741-2754. doi: 10.1002/ehf2.13344. Epub 2021 May 2. PMID 33934542
- [Derived] Averbuch T, Lee SF, Mamas MA, Oz UE, Perez R, Connolly SJ, Ko DT, Van Spall HGC. Derivation and validation of a two-variable index to predict 30-day outcomes following heart failure hospitalization. ESC Heart Fail. 2021 Aug;8(4):2690-2697. doi: 10.1002/ehf2.13324. Epub 2021 May 1. PMID 33932113
- [Derived] Van Spall HG, Averbuch T, Lee SF, Oz UE, Mamas MA, Januzzi JL, Ko DT. The LENT index predicts 30 day outcomes following hospitalization for heart failure. ESC Heart Fail. 2021 Feb;8(1):518-526. doi: 10.1002/ehf2.13109. Epub 2020 Dec 2. PMID 33269549
- [Derived] Van Spall HGC, Lee SF, Xie F, Oz UE, Perez R, Mitoff PR, Maingi M, Tjandrawidjaja MC, Heffernan M, Zia MI, Porepa L, Panju M, Thabane L, Graham ID, Haynes RB, Haughton D, Simek KD, Ko DT, Connolly SJ. Effect of Patient-Centered Transitional Care Services on Clinical Outcomes in Patients Hospitalized for Heart Failure: The PACT-HF Randomized Clinical Trial. JAMA. 2019 Feb 26;321(8):753-761. doi: 10.1001/jama.2019.0710. PMID 30806695
- [Derived] Van Spall HGC, Lee SF, Xie F, Ko DT, Thabane L, Ibrahim Q, Mitoff PR, Heffernan M, Maingi M, Tjandrawidjaja MC, Zia MI, Panju M, Perez R, Simek KD, Porepa L, Graham ID, Haynes RB, Haughton D, Connolly SJ. Knowledge to action: Rationale and design of the Patient-Centered Care Transitions in Heart Failure (PACT-HF) stepped wedge cluster randomized trial. Am Heart J. 2018 May;199:75-82. doi: 10.1016/j.ahj.2017.12.013. Epub 2017 Dec 27. PMID 29754670